CLINICAL TRIAL: NCT03343418
Title: Placebo-Controlled, Randomized, Double-Blind Trial of Prophylactic Desmopressin in Heart Valve Surgery
Brief Title: Effects of Prophylactic Desmopressin on Blood Coagulation Parameters in Heart Valve Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto do Coracao (Other Government)
Responsible Party: Principal Investigator, Filomena R B G Galas, Associate Professor, Instituto do Coracao
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3962.13.087
Record Dates: First submitted 2017-10-10; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: C.Surgical Procedure; Cardiac; Blood Coagulation Disorders
Keywords: Bleeding; Valve Cardiac Surgery; Desmopressin
MeSH Terms: conditions — Blood Coagulation Disorders; Hemorrhage | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- desmopressin (Active Comparator): Patients randomized to this group receive desmopressin 0,3 microgram.kg-1 as an intravenous infusion given during 20 min.
  Interventions: Drug: Desmopressin
- Placebo (Placebo Comparator): Patients randomized to the control group will receive the infusion of 100 mL 0.9% saline (SF0,9%).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desmopressin — Desmopressin is to be administered as an intravenous infusion after discontinuation of cardiopulmonary bypass and administration of protamine. Subjects are to be given desmopressin 0,3 microgram.kg-1. After desmopressin infusion, bleeding treatment will follow the predefined standardized treatment regimen.
  Arms: desmopressin
Drug: Placebo — 0.9% saline is to be administered as an intravenous infusion after discontinuation of cardiopulmonary bypass and administration of protamine. Patients randomized to the control group will receive the infusion of 100 milliliters (mL) 0.9% saline (SF0,9%). After 0.9% saline infusion, bleeding treatment will follow the predefined standardized treatment regimen.
  Arms: Placebo

SUMMARY:
The purpose of this study is evaluate the effect of prophylactic desmopressin on blood coagulation parameters and postoperative bleeding in patients undergoing valve cardiac surgery with cardiopulmonary bypass.

DETAILED DESCRIPTION:
Patients with important valve disorders may evaluate with coagulopathy induced by mechanical effects (valvular stenosis or valvular insufficiency). Furthermore, frequently is required prophylactic use of antiplatelet drugs due to myocardial remodeling and antiarrhythmic conditions that may be associated. Patients with severe aortic stenosis may also acquired von Willebrand disease type 2A due to proteolysis of vonWillebrand factor. Despite of this, the treatment of valve disorders often requires cardiac surgery with cardiopulmonary bypass. On average 50 to 60% of patients undergoing cardiac surgery receive blood tranfusions. Blood cell transfusion is an independent risk factor for increased morbidity and mortality in critically ill patients. The use of desmopressin seems beneficial only in patients with congenital or acquired platelet dysfunction. In general population, such use is not validated due to inconclusive results of researches.

ELIGIBILITY:
Inclusion Criteria:

* Valve cardiac surgery with cardiopulmonary bypass.
* Written informed consent

Exclusion Criteria:

* Reoperative valve surgery
* Hematocrit < 35%
* Ventricular dysfunction (EF < 40%)
* Infection
* Body mass index > 35
* Renal impairment (Creatinin > 2mg/dL)
* Antiplatelet administration within 10 days preceding study surgery
* Participation in another interventional clinical study within 30 days
* Known or suspected hypersensitivity to the desmopressin
* Coagulopathy (INR > 1.5)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Change in coagulation parameters | Coagulation parameters will be performed: T0: preoperative period; T1 - 2 hours after desmopressin or placebo administration; T2 - 24 hours after desmopressin or placebo administration
  Laboratory variables: Activated partial thromboplastin time [(aPTT) seconds], prothrombin time [(PT) seconds], haematocrit (%), haemoglobin(g/dl), fibrinogen(mg/dL), D dimer (ng/L), factor VIII(%), Von Willebrand factor(%), ROTEM [(INTEM, EXTEM, FIBTEM) Clotting Time (CT) and Clot Formation Time (CFT) seconds, alpha angle (α º), Maximum Clot Firmness (MCF) mm ] and platelets aggregation (%)
Postoperative blood loss | 48 hours
  Total chest tube drainage (mL) starting immediately after closure of the chest in the operating theater until 48 hours

SECONDARY OUTCOMES:
Blood transfusion | 30 days
  Number of units of red blood cells, fresh frozen plasma,platelets, cryoprecipitate in the operating theater and ICU
Reoperation for bleeding | 30 days
Duration of Mechanical ventilation | 30 days
Length of vasoactive drugs | 30 days
Length of ICU stay | 30 days
Clinical complications - renal failure, infection, myocardial ischemia, stroke | 30 days
Length of hospital stay | 30 days
Mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Incor - Heart Institute - University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Galas FR, de Almeida JP, Fukushima JT, Vincent JL, Osawa EA, Zeferino S, Camara L, Guimaraes VA, Jatene MB, Hajjar LA. Hemostatic effects of fibrinogen concentrate compared with cryoprecipitate in children after cardiac surgery: a randomized pilot trial. J Thorac Cardiovasc Surg. 2014 Oct;148(4):1647-55. doi: 10.1016/j.jtcvs.2014.04.029. Epub 2014 Apr 18. PMID 24951020